CLINICAL TRIAL: NCT06012344
Title: The Effectiveness of Muscle Energy Technique and Hamstring Nordic Lower in Hamstring Tightness Amongst Young Athletes of Pakistan
Brief Title: Muscle Energy Technique and Hamstring Nordic Lower for Hamstring Tightness in Young Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bhutta001
Record Dates: First submitted 2023-07-01; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Hamstring Tightness; Athletic Injuries; Athletic Performance
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: This triple-blinded, randomized clinical trial employed a five-phase crossover design to evaluate the effects of post-isometric relaxation, post-facilitation stretch, and hamstring Nordic lower exercises on hamstring function and athletic performance in young athletes. Participants were randomly assigned to treatment groups in Phase I, followed by washout periods in Phases II and IV. In Phase III, participants switched treatments to ensure exposure to all interventions. Outcome measures included hamstring flexibility, lower limb power, speed and acceleration, hamstring strength, and agility. The study utilized triple-blinding and randomization to minimize biases. The findings will guide practitioners and coaches in optimizing training and rehabilitation strategies for young athletes. In conclusion, this trial provides valuable insights into the effects of different treatments on hamstring function and athletic performance, benefiting athletes and enhancing performance outcomes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This triple-blinded randomized clinical trial ensured masking of participants, physiotherapists, assessors, and the principal investigator. Participants were unaware of their assigned treatment, as treatments were standardized and shared similar characteristics. Physiotherapists were trained to deliver treatments without disclosing specific interventions. Assessors remained blinded to treatment assignments, conducting outcome assessments independently. The principal investigator had no knowledge of treatment allocations to maintain objectivity. Implementing triple-blinding enhanced the study's internal validity, minimizing biases and improving the reliability of the results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): 20 participant randomly allocated they were administered in first phase with post facilitation stretch , 3rd phase with post isometric relaxation and then in 5th phase hamstring Nordic lower
  Interventions: Other: post facilitation stretch; Other: post isometric relaxation; Other: hamstring nordic lower
- Group B (Experimental): 20 participant randomly allocated they were administered in first phase with post isometric relaxation 3rd phase with hamstring Nordic lower and then in 5th phase post facilitation stretch
  Interventions: Other: post facilitation stretch; Other: post isometric relaxation; Other: hamstring nordic lower
- Group C (Experimental): 20 participant randomly allocated they were administered in first phase hamstring Nordic lower 3rd phase with post facilitation stretch and then in 5th phase post isometric relaxation
  Interventions: Other: post facilitation stretch; Other: post isometric relaxation; Other: hamstring nordic lower

INTERVENTIONS:
Other: post facilitation stretch — PFS Post-Facilitation Stretch Participants in this arm received the intervention of post-facilitation stretch technique. Post-facilitation stretch involves the application of manual stretching techniques to the targeted muscles after a facilitation phase, which aims to enhance muscle extensibility. The participants underwent a standardized post-facilitation stretch protocol focusing on the hamstring muscles.
  Other Names: Muscle energy technique type II
Other: post isometric relaxation — Participants in this arm of the study received the intervention of post-isometric relaxation technique. Post-isometric relaxation involves the application of isometric contraction followed by a relaxation phase to promote muscle lengthening and improve flexibility. The participants underwent a standardized post-isometric relaxation protocol targeting the hamstring muscles.
  Other Names: Muscle energy technique type I
Other: hamstring nordic lower — Participants in this arm received the intervention of hamstring Nordic lower exercise. The hamstring Nordic lower exercise is a challenging eccentric exercise that specifically targets the hamstring muscles. Participants performed the exercise under supervision and followed a standardized protocol for the number of repetitions, sets, and rest intervals.

SUMMARY:
the study aims to assess the efficacy of two interventions, namely the muscle energy technique and the hamstring Nordic lower exercise, in addressing hamstring tightness among young athletes in Pakistan.

DETAILED DESCRIPTION:
Title: The Effectiveness of Muscle Energy Technique and Hamstring Nordic Lower Exercise in Managing Hamstring Tightness Among Young Athletes of Pakistan

Objective:

The primary objective of this study is to investigate the effectiveness of two interventions, the muscle energy technique and the hamstring Nordic lower exercise, in managing hamstring tightness among young athletes from Pakistan.

Background:

Hamstring tightness is a prevalent issue among athletes, which can lead to reduced flexibility, increased risk of injury, and impaired athletic performance. The muscle energy technique is a manual therapy approach that involves active muscle contractions and stretches to improve muscle flexibility and restore normal range of motion. Conversely, the hamstring Nordic lower exercise is a specific eccentric strengthening exercise that targets the hamstring muscles and aims to improve their lengthening capacity.

Study Design:

A randomized controlled trial will be conducted to evaluate the efficacy of the two interventions. Young athletes from Pakistan with hamstring tightness will be recruited as participants. They will be randomly assigned to one of two intervention groups: the muscle energy technique group or the hamstring Nordic lower exercise group. The interventions will be administered by trained healthcare professionals under supervision, following a specific duration and frequency.

Outcome Measures:

The primary outcome measure of interest in this study is the change in hamstring tightness. The measurement tools used to assess this outcome will be reliable and validated. Baseline assessments will be conducted before the intervention period, and post-intervention assessments will take place immediately after the intervention period.

Secondary outcome measures may include improvements in hamstring flexibility, functional performance, and self-reported symptoms related to hamstring tightness. These secondary measures will provide a comprehensive evaluation of the effectiveness of each intervention.

Data Analysis:

Data will be analyzed using appropriate statistical methods. The outcomes between the two intervention groups will be compared to determine the relative effectiveness of the muscle energy technique and the hamstring Nordic lower exercise in managing hamstring tightness.

Implications:

The findings of this research will offer valuable insights into the most suitable intervention for managing hamstring tightness among young athletes in Pakistan. This information can contribute to the development of targeted rehabilitation protocols and injury prevention strategies in this specific population. Furthermore, the results may also have broader implications for similar populations of athletes globally who face similar issues with hamstring tightness.

Conclusion:

By evaluating the effectiveness of the muscle energy technique and the hamstring Nordic lower exercise, this study aims to contribute to the advancement of evidence-based interventions for managing hamstring tightness. The results will be disseminated through scientific publications and presented at relevant conferences to ensure that the knowledge reaches the appropriate healthcare professionals, coaches, and athletes.

ELIGIBILITY:
Inclusion Criteria:

* Athletes with Hamstring tightness
* Both male and female will be included.
* Athletes ages form 18 to 25 years
* athletes having SLR <110˚

Exclusion Criteria:

* Athletes having hamstring injuries
* Patients having painful SLR
* Other orthopedic conditions like LBP,
* Athletes with any deformity
* Recent surgery

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
hamstring nordic Lower test | phase 1 at baseline
  The hamstring Nordic lower test is a functional assessment that evaluates the eccentric strength and endurance of the hamstring muscles. During the test, the participant kneels with the ankles secured and gradually lowers their upper body towards the ground while maintaining control. The goal is to use the hamstrings to control the descent and return to the starting position. This test specifically targets the eccentric contraction of the hamstrings, which is crucial for deceleration, change of direction, and injury prevention. By assessing hamstring strength and endurance, the test can identify weaknesses or imbalances that may increase the risk of hamstring injuries.
hamstring nordic Lower test | phase 1 post intervention 14th day
  The hamstring Nordic lower test is a functional assessment that evaluates the eccentric strength and endurance of the hamstring muscles. During the test, the participant kneels with the ankles secured and gradually lowers their upper body towards the ground while maintaining control. The goal is to use the hamstrings to control the descent and return to the starting position. This test specifically targets the eccentric contraction of the hamstrings, which is crucial for deceleration, change of direction, and injury prevention. By assessing hamstring strength and endurance, the test can identify weaknesses or imbalances that may increase the risk of hamstring injuries.
hamstring nordic Lower test | phase 2 at baseline (after 4 week of washout period)
  The hamstring Nordic lower test is a functional assessment that evaluates the eccentric strength and endurance of the hamstring muscles. During the test, the participant kneels with the ankles secured and gradually lowers their upper body towards the ground while maintaining control. The goal is to use the hamstrings to control the descent and return to the starting position. This test specifically targets the eccentric contraction of the hamstrings, which is crucial for deceleration, change of direction, and injury prevention. By assessing hamstring strength and endurance, the test can identify weaknesses or imbalances that may increase the risk of hamstring injuries.
hamstring nordic Lower test | phase 2 post intervention 14th day
  The hamstring Nordic lower test is a functional assessment that evaluates the eccentric strength and endurance of the hamstring muscles. During the test, the participant kneels with the ankles secured and gradually lowers their upper body towards the ground while maintaining control. The goal is to use the hamstrings to control the descent and return to the starting position. This test specifically targets the eccentric contraction of the hamstrings, which is crucial for deceleration, change of direction, and injury prevention. By assessing hamstring strength and endurance, the test can identify weaknesses or imbalances that may increase the risk of hamstring injuries.
hamstring nordic Lower test | phase 3 at baseline (after 4 week of washout period)
  The hamstring Nordic lower test is a functional assessment that evaluates the eccentric strength and endurance of the hamstring muscles. During the test, the participant kneels with the ankles secured and gradually lowers their upper body towards the ground while maintaining control. The goal is to use the hamstrings to control the descent and return to the starting position. This test specifically targets the eccentric contraction of the hamstrings, which is crucial for deceleration, change of direction, and injury prevention. By assessing hamstring strength and endurance, the test can identify weaknesses or imbalances that may increase the risk of hamstring injuries.
hamstring nordic Lower test | phase 3 post intervention 14th day
  The hamstring Nordic lower test is a functional assessment that evaluates the eccentric strength and endurance of the hamstring muscles. During the test, the participant kneels with the ankles secured and gradually lowers their upper body towards the ground while maintaining control. The goal is to use the hamstrings to control the descent and return to the starting position. This test specifically targets the eccentric contraction of the hamstrings, which is crucial for deceleration, change of direction, and injury prevention. By assessing hamstring strength and endurance, the test can identify weaknesses or imbalances that may increase the risk of hamstring injuries.
100 meter sprint | phase 1 at baseline
  The 100-meter sprint is typically performed in a single continuous effort, with athletes starting from a stationary position and sprinting as fast as possible to reach the finish line.
100 meter sprint | phase 1 post intervention 14th day
  The 100-meter sprint is typically performed in a single continuous effort, with athletes starting from a stationary position and sprinting as fast as possible to reach the finish line.
100 meter sprint | phase 2 at baseline (after 4 week of washout period)
  The 100-meter sprint is typically performed in a single continuous effort, with athletes starting from a stationary position and sprinting as fast as possible to reach the finish line.
100 meter sprint | phase 2 post intervention 14th day
  The 100-meter sprint is typically performed in a single continuous effort, with athletes starting from a stationary position and sprinting as fast as possible to reach the finish line.
100 meter sprint | phase 3 at baseline (after 4 week of washout period)
  The 100-meter sprint is typically performed in a single continuous effort, with athletes starting from a stationary position and sprinting as fast as possible to reach the finish line.
100 meter sprint | phase 3 post intervention 14th day
  The 100-meter sprint is typically performed in a single continuous effort, with athletes starting from a stationary position and sprinting as fast as possible to reach the finish line.
agility run test | phase 1 at baseline
  The agility run test is commonly used in sports that require quick changes of direction, such as soccer, basketball, tennis, and football. It helps to evaluate an athlete's ability to accelerate, decelerate, and change direction efficiently, which are crucial skills for success in these sports.
agility run test | phase 1 post intervention 14th day
  The agility run test is commonly used in sports that require quick changes of direction, such as soccer, basketball, tennis, and football. It helps to evaluate an athlete's ability to accelerate, decelerate, and change direction efficiently, which are crucial skills for success in these sports.
agility run test | phase 2 at baseline (after 4 week of washout period)
  The agility run test is commonly used in sports that require quick changes of direction, such as soccer, basketball, tennis, and football. It helps to evaluate an athlete's ability to accelerate, decelerate, and change direction efficiently, which are crucial skills for success in these sports.
agility run test | phase 2 post intervention 14th day
  The agility run test is commonly used in sports that require quick changes of direction, such as soccer, basketball, tennis, and football. It helps to evaluate an athlete's ability to accelerate, decelerate, and change direction efficiently, which are crucial skills for success in these sports.
agility run test | phase 3 at baseline (after 4 week of washout period)
  The agility run test is commonly used in sports that require quick changes of direction, such as soccer, basketball, tennis, and football. It helps to evaluate an athlete's ability to accelerate, decelerate, and change direction efficiently, which are crucial skills for success in these sports.
agility run test | phase 3 post intervention 14th day
  The agility run test is commonly used in sports that require quick changes of direction, such as soccer, basketball, tennis, and football. It helps to evaluate an athlete's ability to accelerate, decelerate, and change direction efficiently, which are crucial skills for success in these sports.
vertical jump | phase 1 at baseline
  By assessing the vertical jump performance, the test indirectly provides insights into the strength and power of the lower body muscles, including the hamstrings. A strong and well-functioning hamstring muscle group is crucial for generating force during the jump and contributing to the overall jump height.
vertical jump | phase 1 post intervention 14th day
  By assessing the vertical jump performance, the test indirectly provides insights into the strength and power of the lower body muscles, including the hamstrings. A strong and well-functioning hamstring muscle group is crucial for generating force during the jump and contributing to the overall jump height.
vertical jump | phase 2 at baseline (after 4 week of washout period)
  By assessing the vertical jump performance, the test indirectly provides insights into the strength and power of the lower body muscles, including the hamstrings. A strong and well-functioning hamstring muscle group is crucial for generating force during the jump and contributing to the overall jump height.
vertical jump | phase 2 post intervention 14th day
  By assessing the vertical jump performance, the test indirectly provides insights into the strength and power of the lower body muscles, including the hamstrings. A strong and well-functioning hamstring muscle group is crucial for generating force during the jump and contributing to the overall jump height.
vertical jump | phase 3 at baseline (after 4 week of washout period)
  By assessing the vertical jump performance, the test indirectly provides insights into the strength and power of the lower body muscles, including the hamstrings. A strong and well-functioning hamstring muscle group is crucial for generating force during the jump and contributing to the overall jump height.
vertical jump | phase 3 post intervention 14th day
  By assessing the vertical jump performance, the test indirectly provides insights into the strength and power of the lower body muscles, including the hamstrings. A strong and well-functioning hamstring muscle group is crucial for generating force during the jump and contributing to the overall jump height.
YMCA sit & reach box | phase 1 at baseline
  The YMCA sit and reach box is a commonly used tool to measure and assess hamstring and lower back flexibility. It consists of a box or platform with a measuring scale and a sliding panel. The participant sits with their legs extended, placing their feet against the box. They then reach forward with both hands, sliding the panel as far as possible along the measuring scale while keeping their knees straight. The distance reached is recorded as the measurement of flexibility. The YMCA sit and reach test provides an objective measurement of hamstring and lower back flexibility and is widely used in research, fitness testing, and clinical assessments. It is a simple and practical tool to evaluate an individual's flexibility level and monitor changes over time.
YMCA sit & reach box | phase 1 post intervention 14th day
  The YMCA sit and reach box is a commonly used tool to measure and assess hamstring and lower back flexibility. It consists of a box or platform with a measuring scale and a sliding panel. The participant sits with their legs extended, placing their feet against the box. They then reach forward with both hands, sliding the panel as far as possible along the measuring scale while keeping their knees straight. The distance reached is recorded as the measurement of flexibility. The YMCA sit and reach test provides an objective measurement of hamstring and lower back flexibility and is widely used in research, fitness testing, and clinical assessments. It is a simple and practical tool to evaluate an individual's flexibility level and monitor changes over time.
YMCA sit & reach box | phase 2 at baseline (after 4 week of washout period)
  The YMCA sit and reach box is a commonly used tool to measure and assess hamstring and lower back flexibility. It consists of a box or platform with a measuring scale and a sliding panel. The participant sits with their legs extended, placing their feet against the box. They then reach forward with both hands, sliding the panel as far as possible along the measuring scale while keeping their knees straight. The distance reached is recorded as the measurement of flexibility. The YMCA sit and reach test provides an objective measurement of hamstring and lower back flexibility and is widely used in research, fitness testing, and clinical assessments. It is a simple and practical tool to evaluate an individual's flexibility level and monitor changes over time.
YMCA sit & reach box | phase 2 post intervention 14th day
  The YMCA sit and reach box is a commonly used tool to measure and assess hamstring and lower back flexibility. It consists of a box or platform with a measuring scale and a sliding panel. The participant sits with their legs extended, placing their feet against the box. They then reach forward with both hands, sliding the panel as far as possible along the measuring scale while keeping their knees straight. The distance reached is recorded as the measurement of flexibility. The YMCA sit and reach test provides an objective measurement of hamstring and lower back flexibility and is widely used in research, fitness testing, and clinical assessments. It is a simple and practical tool to evaluate an individual's flexibility level and monitor changes over time.
YMCA sit & reach box | phase 3 at baseline (after 4 week of washout period)
  The YMCA sit and reach box is a commonly used tool to measure and assess hamstring and lower back flexibility. It consists of a box or platform with a measuring scale and a sliding panel. The participant sits with their legs extended, placing their feet against the box. They then reach forward with both hands, sliding the panel as far as possible along the measuring scale while keeping their knees straight. The distance reached is recorded as the measurement of flexibility. The YMCA sit and reach test provides an objective measurement of hamstring and lower back flexibility and is widely used in research, fitness testing, and clinical assessments. It is a simple and practical tool to evaluate an individual's flexibility level and monitor changes over time.
YMCA sit & reach box | phase 3 post intervention 14th day
  The YMCA sit and reach box is a commonly used tool to measure and assess hamstring and lower back flexibility. It consists of a box or platform with a measuring scale and a sliding panel. The participant sits with their legs extended, placing their feet against the box. They then reach forward with both hands, sliding the panel as far as possible along the measuring scale while keeping their knees straight. The distance reached is recorded as the measurement of flexibility. The YMCA sit and reach test provides an objective measurement of hamstring and lower back flexibility and is widely used in research, fitness testing, and clinical assessments. It is a simple and practical tool to evaluate an individual's flexibility level and monitor changes over time.

SECONDARY OUTCOMES:
Hamstring Eccentric Testing Questionnaire | phase 1 at baseline
  This questionnaire aims to gather information about athlete experiences and perceptions related to hamstring eccentric testing. The purpose of the questionnaire is to gather valuable insights that can contribute to the development and improvement of hamstring eccentric testing protocols. athlete participation and honest responses are greatly appreciated.
Hamstring Eccentric Testing Questionnaire | phase 1 post intervention 14th day
  This questionnaire aims to gather information about athlete experiences and perceptions related to hamstring eccentric testing. The purpose of the questionnaire is to gather valuable insights that can contribute to the development and improvement of hamstring eccentric testing protocols. athlete participation and honest responses are greatly appreciated.
Hamstring Eccentric Testing Questionnaire | phase 2 at baseline (after 4 week of washout period)
  This questionnaire aims to gather information about athlete experiences and perceptions related to hamstring eccentric testing. The purpose of the questionnaire is to gather valuable insights that can contribute to the development and improvement of hamstring eccentric testing protocols. athlete participation and honest responses are greatly appreciated.
Hamstring Eccentric Testing Questionnaire | phase 2 post intervention 14th day
  This questionnaire aims to gather information about athlete experiences and perceptions related to hamstring eccentric testing. The purpose of the questionnaire is to gather valuable insights that can contribute to the development and improvement of hamstring eccentric testing protocols. athlete participation and honest responses are greatly appreciated.
Hamstring Eccentric Testing Questionnaire | phase 3 at baseline (after 4 week of washout period)
  This questionnaire aims to gather information about athlete experiences and perceptions related to hamstring eccentric testing. The purpose of the questionnaire is to gather valuable insights that can contribute to the development and improvement of hamstring eccentric testing protocols. athlete participation and honest responses are greatly appreciated.
Hamstring Eccentric Testing Questionnaire | phase 3 post intervention 14th day
  This questionnaire aims to gather information about athlete experiences and perceptions related to hamstring eccentric testing. The purpose of the questionnaire is to gather valuable insights that can contribute to the development and improvement of hamstring eccentric testing protocols. athlete participation and honest responses are greatly appreciated.

CONTACTS AND LOCATIONS:
Overall Officials: waqar Ahmed Awan, Ph.D, Study Director — HERF
Locations (1):
- Health Educaiton & research Foundation, Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
URL: http://herf.org.pk